CLINICAL TRIAL: NCT02343497
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group Design, Monocentric Study on Lipid-lowering Effects of an Astaxanthin Supplement in Volunteers With Mild Dyslipidemia
Brief Title: Lipid-lowering Effects of an Astaxanthin Supplement in Volunteers With Mild Dyslipidaemia
Acronym: LLAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajinomoto Foods Europe SAS (Industry)
Collaborators: Institut Polytechnique LaSalle Beauvais (Other); Naturalpha (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2014-A00198-39
Record Dates: First submitted 2015-01-08; First posted 2015-01-22 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Astaxanthin (Experimental): Astaxanthin supplement from Phaffia rhodozyma, 6mg in lipid capsules, 2 caps per day, duration 12 weeks
  Interventions: Dietary Supplement: Astaxanthin
- Placebo (Placebo Comparator): filling agent, in lipid capsules, 2 caps per day, duration 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin
  Arms: Astaxanthin
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether astaxanthin supplementation can impact triglyceride plasmatic concentrations in volunteers presenting mild dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

To be fulfilled at V0:

1. Male and female volunteers, able to read and write, aged from 18 to 60 years inclusive at time of screening.
2. Smokers and no smokers.
3. Subject with a good physical condition confirmed based on the subject's interview and the clinical exam performed by the investigator.
4. Subject with a Body Mass Index (BMI) ≥ 18,5 and < 35 kg/m².
5. Written informed consent provided prior to screening, after receiving and understanding the subject information.
6. Stable body weight (< 3% variation) within the last 3 months prior to screening.
7. Subject registered with the French Social Security, in agreement with the French law on biomedical experimentation.

   To be fulfilled before V1, randomization visit:
8. Subject with fasting triglyceride concentration ≥ 1.2 and < 4 g/l.
9. Subject with fasting serum LDL-cholesterol ≤ 2.2 g/l.

Exclusion Criteria:

To be fulfilled at V0:

1. Subject taking lipid altering drug therapy within 6 weeks prior to screening. Also excluded are supplements known to have significant lipid altering effects, such as:

   * Phytosterols or phytostanols,
   * Red yeast rice extract (Monascus purpureus),
   * Beta-glucans,
   * Omega-3 fatty acids (alpha-linolenic, docosahexaenoic and eicosapentaenoic),
2. Subject using the following medications: systemic corticosteroids (nasal and inhaled corticosteroids are permitted), orlistat, bile acid resins, prescription omega-3 fatty acids, cyclical or non continuous hormone therapy (estrogen or testosterone) excepted stable oestroprogestative or progestative contraception i.e. started at least three months preceding the screening visit.
3. Intake of oestroprogestative or progestative contraception started within less than three months preceding the screening visit.
4. Subject taking antioxidant agents or vitamins within 6 weeks prior to screening.
5. Subject taking astaxanthin-rich foods (red fish and seafood, mostly) or supplements (including krill).
6. Subject following any special diet including, but not limited to liquid, high or low protein, raw food, vegetarian or vegan, etc.
7. Subject with any sensitivity or allergy to any of the products used in this clinical trial.
8. Subject that consume more than three (3) units of alcoholic beverage daily. For the purpose of this study, a unit of alcohol is defined as 400 ml of beer, 200 ml of wine or 50 ml of hard spirits.
9. Subject with known human immunodeficiency virus (HIV) seropositivity.
10. Women who are pregnant or breastfeeding, or planning a pregnancy during the duration of the study.
11. Female subject without efficient contraceptive method: hormonal contraception (including patch, contraceptive ring, etc.), intra-uterine device or other mechanical contraception method (condom or diaphragm) or spermicide for all the duration of the study.
12. Subject treated for type 1 or type 2 diabetes mellitus.
13. Subject with known cardiovascular disease or stroke, except for conditions that are deemed clinically insignificant by the investigator.
14. Subject with symptomatic hypertension, treated or not.
15. Subject treated by antivitamin K.
16. Subject with history of significant gastrointestinal disease such as severe constipation, diarrhea, malabsorptive disease, inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis) and all kind of gastrointestinal surgery.
17. Subject with thyroid dysfunction or treatment for this pathology.
18. Subject with history of severe psychiatric illness which in the opinion of the investigator would interfere with the optimal participation in the study.
19. Subject with history of cancer within 5 years of screening visit (except for successfully treated basal and squamous cell carcinoma of the skin).
20. Subject with any medical contraindication to blood sampling (anemia, clotting defect).
21. Subject practicing intense physical activity (sport, physical exertion at work).
22. Subject with history of drug abuse.
23. Participation to any other clinical trial simultaneously and/or within 1 month prior to screening.
24. Subject who in the opinion of the investigator have a risk of non-compliance to the study procedures or who are otherwise not appropriate to include in this clinical trial.
25. Subject of legal age unable of giving consent.
26. Subject deprived of liberty by judicial or administrative decision.
27. Subject of legal age under legal protection.
28. Subject having received over 4500 euros for clinical trial participation within the prior year including the indemnity for the present study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
fasting plasma triglycerides | 0, 12 weeks
  g/l

SECONDARY OUTCOMES:
fasting cholesterol | 0, 12 weeks
  total cholesterol (g/l)
fasting HDL-cholesterol | 0, 12 weeks
  g/l
fasting LDL-cholesterol | 0, 12 weeks
  g/l
apolipoprotein A1 | 0, 12 weeks
  g/l
apolipoprotein B | 0, 12 weeks
  g/l
apolipoprotein balance | 0, 12 weeks
  Apolipoprotein B over Apolipoprotein A1 ratio
resting blood pressure | 0, 6, 12 weeks
  triplicate measure
resting heart rate | 0, 6, 12 weeks
fasting glucose | 0, 12 weeks
  g/l
fasting insulin | 0, 12 weeks
  mU/l
homeostatic model assessment to quantify insulin resistance (HOMA-IR) | 0, 12 weeks
  glucose (mg/dl) * insulin(U/l) / 405
fasting adiponectin | 0, 12 weeks
  flow cytometry
fasting leptin | 0, 12 weeks
  flow cytometry
fasting ghrelin | 0, 12 weeks
  flow cytometry
fasting resistin | 0, 12 weeks
  flow cytometry
phosphatidylcholine hydroperoxides | 0, 12 weeks
  HPLC/MS
plasmatic concentrations in astaxanthin | 0, 6, 12 weeks
  HPLC/MS
compliance with study product | 0, 6, 12 weeks
  accountability of returned used/unused caps
adverse events | during the 12 weeks of intervention
  number of subjects with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Nutrition Clinique Naturalpha, Lille, France